CLINICAL TRIAL: NCT05660031
Title: Treatment of the Biceps With Concomitant Supraspinatus Tears: A Multicenter Pragmatic Three-Arm Parallel-Group Randomized Surgical Trial
Brief Title: Treatment of the Biceps With Concomitant Supraspinatus Tears
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: La Tour Hospital (Other)
Responsible Party: Principal Investigator, Dr. Alexandre Lädermann, Orthopaedic Surgeon FMH, Shoulder and Elbow Surgery Traumatology, La Tour Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-00066
Record Dates: First submitted 2022-12-04; First posted 2022-12-21 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Supraspinatus Tear
Keywords: Long head of the biceps; Supraspinatus tear; tenotomy; tenodesis; rotator cuff repair

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Leaving LHB Intact (No Intervention): The long head of the biceps (LHB) will be left intact.
- LHB tenotomy (Experimental): The long head of the biceps (LHB) will be cut at its origin.
  Interventions: Procedure: LHB Tenotomy
- LHB Tenodesis (Experimental): The long head of the biceps (LHB) will be cut at its origin and reattached.
  Interventions: Procedure: LHB Tenodesis

INTERVENTIONS:
Procedure: LHB Tenotomy — Will be performed arthroscopically by cutting the LHB at its origin with arthroscopic scissors
  Arms: LHB tenotomy
Procedure: LHB Tenodesis — "ill be performed arthroscopically with a tenodesis at the top of the articular margin using an onlay technique.
  Arms: LHB Tenodesis

SUMMARY:
The long head of the biceps (LHB) tendon is thought to be a common source of shoulder pain and dysfunction in patients with rotator cuff pathology. Tenotomy and tenodesis have been shown to produce favourable and comparable results in treating LHB lesions, but a controversy still exists regarding the treatment of choice. Some suggest that tenotomy should be reserved for older, low-demand patients, while tenodesis should be performed in younger patients and those who engage in heavy labor. Proponents of tenotomy suggest that this is a technically easy procedure that leads to easy rehabilitation and fast return to activity with a low complication and reoperation rate. However, those who support LHB tenodesis list good preservation of elbow flexion and supination strength, improvement of functional scores, elimination of pain, and avoidance of cosmetic deformity as benefits of the procedure. Alternatively, the LHB can be maintained in the joint without tenodesis or tenotomy. In fact, it has not been clearly shown that LHB tenodesis or tenotomy leads to improved outcomes compared to leaving the biceps tendon intact.

DETAILED DESCRIPTION:
The long head of the biceps (LHB) tendon is thought to be a common source of shoulder pain and dysfunction in patients with rotator cuff pathology.Tenotomy and tenodesis have been shown to produce favourable and comparable results in treating LHB lesions, but a controversy still exists regarding the treatment of choice. Some suggest that tenotomy should be reserved for older, low-demand patients, while tenodesis should be performed in younger patients and those who engage in heavy labor. Proponents of tenotomy suggest that this is a technically easy procedure that leads to easy rehabilitation and fast return to activity with a low complication and reoperation rate. However, those who support LHB tenodesis list good preservation of elbow flexion and supination strength, improvement of functional scores, elimination of pain, and avoidance of cosmetic deformity as benefits of the procedure. Alternatively, the LHB can be maintained in the joint without tenodesis or tenotomy. In fact, it has not been clearly shown that LHB tenodesis or tenotomy leads to improved outcomes compared to leaving the biceps tendon intact. The primary goal of this prospective multicenter randomized study is to evaluate whether LHB tenodesis grants superior post-operative functional outcomes compared to LHB tenotomy or leaving the LHB intact in patients undergoing rotator cuff repair (RCR) for an isolated full-thickness lesion of the supraspinatus. The primary goal of this prospective multicenter randomized study is to evaluate whether LHB tenodesis grants superior post-operative functional outcomes compared to LHB tenotomy or leaving the LHB intact in patients undergoing rotator cuff repair (RCR) for an isolated full-thickness lesion of the supraspinatus. The secondary goals are to determine whether there is a difference in post-operative functional outcomes between the LHB tenotomy group and the Intact LHB group, and if there is a difference in complication rates or patient satisfaction between the three groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient voluntarily consents to participate in the study and has the mental and physical ability to participate in the study, fill out subjective questionnaires, return for follow-up visits, and comply with prescribed post-operative physical therapy.
* Full thickness tear of the supraspinatus tendon
* Intact subscapularis tendon
* Primary rotator cuff repair
* Age 50-80

Exclusion Criteria:

* Previous full thickness biceps tear
* Infection and neuropathic joints
* Known or suspected non-compliance, drug or alcohol abuse
* Patients incapable of judgement or under tutelage
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, contraindication for MRI scan etc.
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Patient declines to participate in study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
ASES score | At 24 post-operative months
  American Shoulder and Elbow Surgeon (ASES) score. From 0 (worst) to 100 (best).

SECONDARY OUTCOMES:
VAS pain | At 24 post-operative months
  Visual analog scale (VAS) pain. From 0 (best) to 10 (worst)
SSV | At 24 post-operative months
  Subjective Shoulder Value (SSV). From 0 (worst) to 100 (best).
LHB score | At 24 post-operative months
  Long head of the biceps (LHB) score. From 0 (worst) to 100 (best).
AFF | At 24 post-operative months
  Anterior Forward Flexion. In degrees. Will be performed with a goniometer by an independent investigator
ER at side | At 24 post-operative months
  External Rotation at the side. In degrees. Will be performed with a goniometer by an independent investigator
IR | At 24 post-operative months
  Internal Rotation to nearest spinal level. Will be performed with a goniometer by an independent investigator
Complications | Within 2 postoperative years
  Any type of post-operative complication
Patient satisfaction | At 24 post-operative months
  Yes or no
Location of the defect (at the foot print | medial cuff failure) | At 6 post-operative month
  Radiographic outcome evaluated using an ultrasound examination.
Status of the biceps tendon (intact | in continuity | defect) | At 6 post-operative month
  Radiographic outcome evaluated using an ultrasound examination.
Signs of anchor displacement and location (lateral | medial row). | At 6 post-operative month
  Radiographic outcome evaluated using an ultrasound examination.
Tendon thickness | At 6 post-operative month
  Radiographic outcome evaluated using an ultrasound examination.
Number of patients with bursitis | At 6 post-operative month
  Radiographic outcome evaluated using an ultrasound examination.
Number of patients with healing of the Supraspinatus tear according to Sugaya classification | At 6 post-operative month
  Radiographic outcome evaluated using an ultrasound examination.
Number of patients with liquid in the bicipital sheath | At 6 post-operative month
  Radiographic outcome evaluated using an ultrasound examination.
Number of patients with hypervascularization of the sheath | At 6 post-operative month
  Radiographic outcome evaluated using an ultrasound examination.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Lädermann, MD, Principal Investigator — La Tour Hospital
Locations (4):
- United States (2):
  - Sports Medicine and Shoulder Surgery, University of Michigan, Ann Arbor, Michigan
  - Oregon Health & Science University, Portland, Oregon
- Group 23 Sports Medicine, Calgary, Alberta, Canada
- la Tour hospital, Meyrin, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No